CLINICAL TRIAL: NCT02417428
Title: Effects of Citrulline Supplementation Combined With Exercise on Muscle Function and Functional Capacity in Older Obese Men and Women
Brief Title: Citrulline Supplementation Combined With Exercise: Effect on Muscle Function in Elderly People (CITEX Study)
Acronym: CITEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: McGill University (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Mylène Aubertin-Leheudre, Professor-Researcher, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N/A with our grant
Record Dates: First submitted 2015-04-02; First posted 2015-04-15 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-06

CONDITIONS: Sarcopenia; Obesity
Keywords: Muscle function; Functional capacity
MeSH Terms: conditions — Sarcopenia; Obesity | interventions — Citrulline; Exercise; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Citrulline (Experimental): Participants that will be randomized in the first arm will be divided in either citrulline plus HIIT (CIT + HIIT or group A) or citrulline alone (CIT or group B).
  Interventions: Dietary Supplement: Citrulline; Other: without exercise
- Placebo (Placebo Comparator): Participants that will be randomized in the second arm will be divided in either placebo plus HIIT (PLA + HIIT or group C) or placebo alone (PLA or group D).
  Interventions: Other: Placebo; Other: without exercise
- Exercise (Experimental): Participant that will be randomized in this arm will have an exercise program (HIIT) added to their respective dietary supplement.
  Interventions: Dietary Supplement: Citrulline; Behavioral: Exercise
- Without exercise (Other): Participant that will be randomized in this arm will not have an exercise program.
  Interventions: Other: Placebo; Behavioral: Exercise

INTERVENTIONS:
Dietary Supplement: Citrulline — Twelve weeks of citrulline oral supplementation will be taken by half of the participants (other are taken a placebo). Citrulline supplementation will be taken orally. Ten grams of citrulline (white powder) will be mixed with a liquid daily. Supplementation will be consumed once at lunch time.
  Arms: Citrulline; Exercise
Other: Placebo — Twelve weeks of oral placebo will be taken by half of the participants. Ten grams of placebo (maltodextrin white powder) will be mixed with a liquid and will be consumed once daily at lunch time.
  Arms: Placebo; Without exercise
Behavioral: Exercise — Participants will also take part in twelve weeks of HIIT (30s at 85% and up of maximal heart rate + 1m30sec at 60-75% of maximal heart rate (HR max). 3 times/ week during 30 continuous minutes. Each period are supervised and monitored using borg scale and polar system.
  Other Names: High intensity interval training (HIIT)
  Arms: Exercise; Without exercise
Other: without exercise — No exercise program will be assigned to participants.
  Arms: Citrulline; Placebo

SUMMARY:
The main objective of this study is to determine if oral supplementation of Citrulline, when combined with HIIT, can produce significant changes in body composition, muscle quality, muscle metabolism and functional capacity in older obese men and women .

The investigators hypothesize that Citrulline combined with HIIT will be more beneficial than HIIT alone which will be more beneficial than citrulline alone which will be more beneficial than placebo alone in obese elderly men and women .

DETAILED DESCRIPTION:
Citrulline is a non-protein amino acid, isolated from watermelon, involved in the urea cycle and an arginine precursor. Participants will take 10g/d of citrulline or placebo (isocaloric).

High intensity interval training (HIIT) is a high intensity aerobic training (30 sec at 85% and up of HRmax + 1min30 at 65-70% of HRmax). they HIIT duration is 30 min/session. HIIT is recognized as beneficial to improve health in human such as Vo2max, body fat or .

Then intervention will be follow during 12 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

1. autonomous (being able to follow the exercise program) and without cognitive impairment (MOCA test ≥21) ;
2. obese status (BMI between 30 and 40 kg / m2 or a waist circumference greater than 102 cm for men and 88 cm for women or fat mass (%; total or androïd or gynoïd) equal or superior to 27% in men and 40% in women;
3. stable weight (± 5 kg) for 6 months;
4. non-smoking and moderate drinkers (max: 15 g/day of alcohol) ;
5. without stroke or history of stroke ;
6. sedentary (less than 2 hours of structured physical activity per week);
7. not being involved in a vigorous exercise program for at least 12 months;
8. can understand French
9. postmenopausal women (without menses since 60 consecutively months).

Exclusion Criteria:

1. to have a metal implant (pacemaker);
2. asthma requiring oral steroid treatment;
3. taking other medication that could affect metabolism or cardiovascular function;
4. taking anticoagulant medication.
5. taking hormonal-replacement therapy (only for women)

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-06; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Improvement in body composition and muscle quality | 12 weeks
  We will determine whether Group A improves more body composition (decreases fat mass (%), increases Leg lean mass index (kg), increases Leg muscle strength (kg)) than group C, B or D.

SECONDARY OUTCOMES:
Exploratory aims: improvements in citrate synthase | 12 weeks
  We will determine whether Group A improves citrate synthase (CS),compared to Group C or B or D.
Exploratory aims:improvements in palmitate oxidation. | 12 weeks
  We will determine whether Group A palmitate oxidation, compared to Group C or B or D.

CONTACTS AND LOCATIONS:
Overall Officials: Mylene Aubertin-Leheudre, PhD, Principal Investigator — Université du Québec a Montréal
Locations (1):
- Universite du Quebec a Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Figueroa A, Alvarez-Alvarado S, Ormsbee MJ, Madzima TA, Campbell JC, Wong A. Impact of L-citrulline supplementation and whole-body vibration training on arterial stiffness and leg muscle function in obese postmenopausal women with high blood pressure. Exp Gerontol. 2015 Mar;63:35-40. doi: 10.1016/j.exger.2015.01.046. Epub 2015 Jan 28. PMID 25636814
- [Background] Moinard C, Nicolis I, Neveux N, Darquy S, Benazeth S, Cynober L. Dose-ranging effects of citrulline administration on plasma amino acids and hormonal patterns in healthy subjects: the Citrudose pharmacokinetic study. Br J Nutr. 2008 Apr;99(4):855-62. doi: 10.1017/S0007114507841110. Epub 2007 Oct 22. PMID 17953788
- [Background] Bahri S, Zerrouk N, Aussel C, Moinard C, Crenn P, Curis E, Chaumeil JC, Cynober L, Sfar S. Citrulline: from metabolism to therapeutic use. Nutrition. 2013 Mar;29(3):479-84. doi: 10.1016/j.nut.2012.07.002. Epub 2012 Sep 28. PMID 23022123
- [Background] Batsis JA, Mackenzie TA, Barre LK, Lopez-Jimenez F, Bartels SJ. Sarcopenia, sarcopenic obesity and mortality in older adults: results from the National Health and Nutrition Examination Survey III. Eur J Clin Nutr. 2014 Sep;68(9):1001-7. doi: 10.1038/ejcn.2014.117. Epub 2014 Jun 25. PMID 24961545
- [Background] Blaum CS, Xue QL, Michelon E, Semba RD, Fried LP. The association between obesity and the frailty syndrome in older women: the Women's Health and Aging Studies. J Am Geriatr Soc. 2005 Jun;53(6):927-34. doi: 10.1111/j.1532-5415.2005.53300.x. PMID 15935013
- [Background] Baumgartner RN. Body composition in healthy aging. Ann N Y Acad Sci. 2000 May;904:437-48. doi: 10.1111/j.1749-6632.2000.tb06498.x. PMID 10865787
- [Background] Cesari M, Pahor M, Lauretani F, Zamboni V, Bandinelli S, Bernabei R, Guralnik JM, Ferrucci L. Skeletal muscle and mortality results from the InCHIANTI Study. J Gerontol A Biol Sci Med Sci. 2009 Mar;64(3):377-84. doi: 10.1093/gerona/gln031. Epub 2009 Jan 30. PMID 19181709
- [Background] Janssen I, Heymsfield SB, Ross R. Low relative skeletal muscle mass (sarcopenia) in older persons is associated with functional impairment and physical disability. J Am Geriatr Soc. 2002 May;50(5):889-96. doi: 10.1046/j.1532-5415.2002.50216.x. PMID 12028177
- [Background] Zamboni M, Mazzali G, Fantin F, Rossi A, Di Francesco V. Sarcopenic obesity: a new category of obesity in the elderly. Nutr Metab Cardiovasc Dis. 2008 Jun;18(5):388-95. doi: 10.1016/j.numecd.2007.10.002. Epub 2008 Apr 18. PMID 18395429
- [Background] Prado CM, Wells JC, Smith SR, Stephan BC, Siervo M. Sarcopenic obesity: A Critical appraisal of the current evidence. Clin Nutr. 2012 Oct;31(5):583-601. doi: 10.1016/j.clnu.2012.06.010. Epub 2012 Jul 17. PMID 22809635
- [Background] Lu Y, Shu H, Zheng Y, Li C, Liu M, Chen Z, He X. Comparison of fat-free mass index and fat mass index in Chinese adults. Eur J Clin Nutr. 2012 Sep;66(9):1004-7. doi: 10.1038/ejcn.2012.86. Epub 2012 Jul 18. PMID 22805496
- [Background] Baumgartner RN, Wayne SJ, Waters DL, Janssen I, Gallagher D, Morley JE. Sarcopenic obesity predicts instrumental activities of daily living disability in the elderly. Obes Res. 2004 Dec;12(12):1995-2004. doi: 10.1038/oby.2004.250. PMID 15687401
- [Background] Rolland Y, Lauwers-Cances V, Cristini C, Abellan van Kan G, Janssen I, Morley JE, Vellas B. Difficulties with physical function associated with obesity, sarcopenia, and sarcopenic-obesity in community-dwelling elderly women: the EPIDOS (EPIDemiologie de l'OSteoporose) Study. Am J Clin Nutr. 2009 Jun;89(6):1895-900. doi: 10.3945/ajcn.2008.26950. Epub 2009 Apr 15. PMID 19369381
- [Background] Vilaca KH, Carneiro JA, Ferriolli E, Lima NK, de Paula FJ, Moriguti JC. Body composition, physical performance and muscle quality of active elderly women. Arch Gerontol Geriatr. 2014 Jul-Aug;59(1):44-8. doi: 10.1016/j.archger.2014.02.004. Epub 2014 Feb 22. PMID 24630334
- [Background] Zoico E, Di Francesco V, Guralnik JM, Mazzali G, Bortolani A, Guariento S, Sergi G, Bosello O, Zamboni M. Physical disability and muscular strength in relation to obesity and different body composition indexes in a sample of healthy elderly women. Int J Obes Relat Metab Disord. 2004 Feb;28(2):234-41. doi: 10.1038/sj.ijo.0802552. PMID 14708033
- [Background] Bouchard DR, Dionne IJ, Brochu M. Sarcopenic/obesity and physical capacity in older men and women: data from the Nutrition as a Determinant of Successful Aging (NuAge)-the Quebec longitudinal Study. Obesity (Silver Spring). 2009 Nov;17(11):2082-8. doi: 10.1038/oby.2009.109. Epub 2009 Apr 16. PMID 19373219
- [Background] Dominguez LJ, Barbagallo M. The cardiometabolic syndrome and sarcopenic obesity in older persons. J Cardiometab Syndr. 2007 Summer;2(3):183-9. doi: 10.1111/j.1559-4564.2007.06673.x. PMID 17786082
- [Background] Barbat-Artigas S, Filion ME, Plouffe S, Aubertin-Leheudre M. Muscle quality as a potential explanation of the metabolically healthy but obese and sarcopenic obese paradoxes. Metab Syndr Relat Disord. 2012 Apr;10(2):117-22. doi: 10.1089/met.2011.0092. Epub 2011 Dec 19. PMID 22182254
- [Background] Hepple RT. Muscle atrophy is not always sarcopenia. J Appl Physiol (1985). 2012 Aug 15;113(4):677-9. doi: 10.1152/japplphysiol.00304.2012. Epub 2012 Apr 19. No abstract available. PMID 22518833
- [Background] Gouspillou G, Sgarioto N, Kapchinsky S, Purves-Smith F, Norris B, Pion CH, Barbat-Artigas S, Lemieux F, Taivassalo T, Morais JA, Aubertin-Leheudre M, Hepple RT. Increased sensitivity to mitochondrial permeability transition and myonuclear translocation of endonuclease G in atrophied muscle of physically active older humans. FASEB J. 2014 Apr;28(4):1621-33. doi: 10.1096/fj.13-242750. Epub 2013 Dec 26. PMID 24371120
- [Background] Picard M, Ritchie D, Wright KJ, Romestaing C, Thomas MM, Rowan SL, Taivassalo T, Hepple RT. Mitochondrial functional impairment with aging is exaggerated in isolated mitochondria compared to permeabilized myofibers. Aging Cell. 2010 Dec;9(6):1032-46. doi: 10.1111/j.1474-9726.2010.00628.x. PMID 20849523
- [Background] Picard M, Ritchie D, Thomas MM, Wright KJ, Hepple RT. Alterations in intrinsic mitochondrial function with aging are fiber type-specific and do not explain differential atrophy between muscles. Aging Cell. 2011 Dec;10(6):1047-55. doi: 10.1111/j.1474-9726.2011.00745.x. PMID 21933339
- [Background] Chabi B, Ljubicic V, Menzies KJ, Huang JH, Saleem A, Hood DA. Mitochondrial function and apoptotic susceptibility in aging skeletal muscle. Aging Cell. 2008 Jan;7(1):2-12. doi: 10.1111/j.1474-9726.2007.00347.x. Epub 2007 Nov 19. PMID 18028258
- [Background] Coen PM, Jubrias SA, Distefano G, Amati F, Mackey DC, Glynn NW, Manini TM, Wohlgemuth SE, Leeuwenburgh C, Cummings SR, Newman AB, Ferrucci L, Toledo FG, Shankland E, Conley KE, Goodpaster BH. Skeletal muscle mitochondrial energetics are associated with maximal aerobic capacity and walking speed in older adults. J Gerontol A Biol Sci Med Sci. 2013 Apr;68(4):447-55. doi: 10.1093/gerona/gls196. Epub 2012 Oct 9. PMID 23051977
- [Background] Conley KE, Esselman PC, Jubrias SA, Cress ME, Inglin B, Mogadam C, Schoene RB. Ageing, muscle properties and maximal O(2) uptake rate in humans. J Physiol. 2000 Jul 1;526 Pt 1(Pt 1):211-7. doi: 10.1111/j.1469-7793.2000.00211.x. PMID 10878113
- [Background] Hagen JL, Krause DJ, Baker DJ, Fu MH, Tarnopolsky MA, Hepple RT. Skeletal muscle aging in F344BN F1-hybrid rats: I. Mitochondrial dysfunction contributes to the age-associated reduction in VO2max. J Gerontol A Biol Sci Med Sci. 2004 Nov;59(11):1099-110. doi: 10.1093/gerona/59.11.1099. PMID 15602055
- [Background] Trounce I, Byrne E, Marzuki S. Decline in skeletal muscle mitochondrial respiratory chain function: possible factor in ageing. Lancet. 1989 Mar 25;1(8639):637-9. doi: 10.1016/s0140-6736(89)92143-0. PMID 2564459
- [Background] Rooyackers OE, Adey DB, Ades PA, Nair KS. Effect of age on in vivo rates of mitochondrial protein synthesis in human skeletal muscle. Proc Natl Acad Sci U S A. 1996 Dec 24;93(26):15364-9. doi: 10.1073/pnas.93.26.15364. PMID 8986817
- [Background] Short KR, Bigelow ML, Kahl J, Singh R, Coenen-Schimke J, Raghavakaimal S, Nair KS. Decline in skeletal muscle mitochondrial function with aging in humans. Proc Natl Acad Sci U S A. 2005 Apr 12;102(15):5618-23. doi: 10.1073/pnas.0501559102. Epub 2005 Mar 30. PMID 15800038
- [Background] Goodpaster BH, Kelley DE, Thaete FL, He J, Ross R. Skeletal muscle attenuation determined by computed tomography is associated with skeletal muscle lipid content. J Appl Physiol (1985). 2000 Jul;89(1):104-10. doi: 10.1152/jappl.2000.89.1.104. PMID 10904041
- [Background] Hulver MW, Berggren JR, Cortright RN, Dudek RW, Thompson RP, Pories WJ, MacDonald KG, Cline GW, Shulman GI, Dohm GL, Houmard JA. Skeletal muscle lipid metabolism with obesity. Am J Physiol Endocrinol Metab. 2003 Apr;284(4):E741-7. doi: 10.1152/ajpendo.00514.2002. Epub 2002 Dec 27. PMID 12626325
- [Background] Cree MG, Newcomer BR, Katsanos CS, Sheffield-Moore M, Chinkes D, Aarsland A, Urban R, Wolfe RR. Intramuscular and liver triglycerides are increased in the elderly. J Clin Endocrinol Metab. 2004 Aug;89(8):3864-71. doi: 10.1210/jc.2003-031986. PMID 15292319
- [Background] Patti ME, Butte AJ, Crunkhorn S, Cusi K, Berria R, Kashyap S, Miyazaki Y, Kohane I, Costello M, Saccone R, Landaker EJ, Goldfine AB, Mun E, DeFronzo R, Finlayson J, Kahn CR, Mandarino LJ. Coordinated reduction of genes of oxidative metabolism in humans with insulin resistance and diabetes: Potential role of PGC1 and NRF1. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8466-71. doi: 10.1073/pnas.1032913100. Epub 2003 Jun 27. PMID 12832613
- [Background] Mootha VK, Lindgren CM, Eriksson KF, Subramanian A, Sihag S, Lehar J, Puigserver P, Carlsson E, Ridderstrale M, Laurila E, Houstis N, Daly MJ, Patterson N, Mesirov JP, Golub TR, Tamayo P, Spiegelman B, Lander ES, Hirschhorn JN, Altshuler D, Groop LC. PGC-1alpha-responsive genes involved in oxidative phosphorylation are coordinately downregulated in human diabetes. Nat Genet. 2003 Jul;34(3):267-73. doi: 10.1038/ng1180. PMID 12808457
- [Background] Kelley DE, Williams KV, Price JC, McKolanis TM, Goodpaster BH, Thaete FL. Plasma fatty acids, adiposity, and variance of skeletal muscle insulin resistance in type 2 diabetes mellitus. J Clin Endocrinol Metab. 2001 Nov;86(11):5412-9. doi: 10.1210/jcem.86.11.8027. PMID 11701715
- [Background] Petersen KF, Befroy D, Dufour S, Dziura J, Ariyan C, Rothman DL, DiPietro L, Cline GW, Shulman GI. Mitochondrial dysfunction in the elderly: possible role in insulin resistance. Science. 2003 May 16;300(5622):1140-2. doi: 10.1126/science.1082889. PMID 12750520
- [Background] Gouspillou G, Sgarioto N, Norris B, Barbat-Artigas S, Aubertin-Leheudre M, Morais JA, Burelle Y, Taivassalo T, Hepple RT. The relationship between muscle fiber type-specific PGC-1alpha content and mitochondrial content varies between rodent models and humans. PLoS One. 2014 Aug 14;9(8):e103044. doi: 10.1371/journal.pone.0103044. eCollection 2014. PMID 25121500
- [Background] Amati F, Dube JJ, Alvarez-Carnero E, Edreira MM, Chomentowski P, Coen PM, Switzer GE, Bickel PE, Stefanovic-Racic M, Toledo FG, Goodpaster BH. Skeletal muscle triglycerides, diacylglycerols, and ceramides in insulin resistance: another paradox in endurance-trained athletes? Diabetes. 2011 Oct;60(10):2588-97. doi: 10.2337/db10-1221. Epub 2011 Aug 26. PMID 21873552
- [Background] Weinberg JM. Lipotoxicity. Kidney Int. 2006 Nov;70(9):1560-6. doi: 10.1038/sj.ki.5001834. Epub 2006 Sep 6. PMID 16955100
- [Background] Choo HJ, Kim JH, Kwon OB, Lee CS, Mun JY, Han SS, Yoon YS, Yoon G, Choi KM, Ko YG. Mitochondria are impaired in the adipocytes of type 2 diabetic mice. Diabetologia. 2006 Apr;49(4):784-91. doi: 10.1007/s00125-006-0170-2. Epub 2006 Feb 25. PMID 16501941
- [Background] Nisoli E, Carruba MO. Emerging aspects of pharmacotherapy for obesity and metabolic syndrome. Pharmacol Res. 2004 Nov;50(5):453-69. doi: 10.1016/j.phrs.2004.02.004. PMID 15458765
- [Background] Chakravarthy MV, Booth FW. Eating, exercise, and "thrifty" genotypes: connecting the dots toward an evolutionary understanding of modern chronic diseases. J Appl Physiol (1985). 2004 Jan;96(1):3-10. doi: 10.1152/japplphysiol.00757.2003. PMID 14660491
- [Background] Golubic R, Martin KR, Ekelund U, Hardy R, Kuh D, Wareham N, Cooper R, Brage S; NSHD scientific and data collection teams. Levels of physical activity among a nationally representative sample of people in early old age: results of objective and self-reported assessments. Int J Behav Nutr Phys Act. 2014 May 3;11:58. doi: 10.1186/1479-5868-11-58. PMID 24885497
- [Background] Coleman KJ, Raynor HR, Mueller DM, Cerny FJ, Dorn JM, Epstein LH. Providing sedentary adults with choices for meeting their walking goals. Prev Med. 1999 May;28(5):510-9. doi: 10.1006/pmed.1998.0471. PMID 10329342
- [Background] Schiffer T, Knicker A, Hoffman U, Harwig B, Hollmann W, Struder HK. Physiological responses to nordic walking, walking and jogging. Eur J Appl Physiol. 2006 Sep;98(1):56-61. doi: 10.1007/s00421-006-0242-5. Epub 2006 Jun 24. PMID 16799817
- [Background] Russ DW, Kent-Braun JA. Is skeletal muscle oxidative capacity decreased in old age? Sports Med. 2004;34(4):221-9. doi: 10.2165/00007256-200434040-00002. PMID 15049714
- [Background] Bruce CR, Thrush AB, Mertz VA, Bezaire V, Chabowski A, Heigenhauser GJ, Dyck DJ. Endurance training in obese humans improves glucose tolerance and mitochondrial fatty acid oxidation and alters muscle lipid content. Am J Physiol Endocrinol Metab. 2006 Jul;291(1):E99-E107. doi: 10.1152/ajpendo.00587.2005. Epub 2006 Feb 7. PMID 16464906
- [Background] Menshikova EV, Ritov VB, Toledo FG, Ferrell RE, Goodpaster BH, Kelley DE. Effects of weight loss and physical activity on skeletal muscle mitochondrial function in obesity. Am J Physiol Endocrinol Metab. 2005 Apr;288(4):E818-25. doi: 10.1152/ajpendo.00322.2004. Epub 2004 Dec 7. PMID 15585590
- [Background] Short KR, Vittone JL, Bigelow ML, Proctor DN, Rizza RA, Coenen-Schimke JM, Nair KS. Impact of aerobic exercise training on age-related changes in insulin sensitivity and muscle oxidative capacity. Diabetes. 2003 Aug;52(8):1888-96. doi: 10.2337/diabetes.52.8.1888. PMID 12882902
- [Background] Henriksson J. Effects of physical training on the metabolism of skeletal muscle. Diabetes Care. 1992 Nov;15(11):1701-11. doi: 10.2337/diacare.15.11.1701. PMID 1468304
- [Background] Holloszy JO, Coyle EF. Adaptations of skeletal muscle to endurance exercise and their metabolic consequences. J Appl Physiol Respir Environ Exerc Physiol. 1984 Apr;56(4):831-8. doi: 10.1152/jappl.1984.56.4.831. PMID 6373687
- [Background] Jobgen WS, Fried SK, Fu WJ, Meininger CJ, Wu G. Regulatory role for the arginine-nitric oxide pathway in metabolism of energy substrates. J Nutr Biochem. 2006 Sep;17(9):571-88. doi: 10.1016/j.jnutbio.2005.12.001. Epub 2006 Jan 9. PMID 16524713
- [Background] Osowska S, Duchemann T, Walrand S, Paillard A, Boirie Y, Cynober L, Moinard C. Citrulline modulates muscle protein metabolism in old malnourished rats. Am J Physiol Endocrinol Metab. 2006 Sep;291(3):E582-6. doi: 10.1152/ajpendo.00398.2005. Epub 2006 Apr 11. PMID 16608884
- [Background] Moinard C, Cynober L. Citrulline: a new player in the control of nitrogen homeostasis. J Nutr. 2007 Jun;137(6 Suppl 2):1621S-1625S. doi: 10.1093/jn/137.6.1621S. PMID 17513438
- [Background] Fujita S, Volpi E. Amino acids and muscle loss with aging. J Nutr. 2006 Jan;136(1 Suppl):277S-80S. doi: 10.1093/jn/136.1.277S. PMID 16365098
- [Background] Le Plenier S, Walrand S, Noirt R, Cynober L, Moinard C. Effects of leucine and citrulline versus non-essential amino acids on muscle protein synthesis in fasted rat: a common activation pathway? Amino Acids. 2012 Sep;43(3):1171-8. doi: 10.1007/s00726-011-1172-z. Epub 2011 Dec 13. PMID 22160257
- [Background] Faure C, Morio B, Chafey P, Le Plenier S, Noirez P, Randrianarison-Huetz V, Cynober L, Aussel C, Moinard C. Citrulline enhances myofibrillar constituents expression of skeletal muscle and induces a switch in muscle energy metabolism in malnourished aged rats. Proteomics. 2013 Jul;13(14):2191-201. doi: 10.1002/pmic.201200262. Epub 2013 Jun 10. PMID 23592530
- [Background] Cynober L, Moinard C, De Bandt JP. The 2009 ESPEN Sir David Cuthbertson. Citrulline: a new major signaling molecule or just another player in the pharmaconutrition game? Clin Nutr. 2010 Oct;29(5):545-51. doi: 10.1016/j.clnu.2010.07.006. Epub 2010 Aug 16. PMID 20719411
- [Background] Joffin N, Jaubert AM, Durant S, Bastin J, De Bandt JP, Cynober L, Moinard C, Coumoul X, Forest C, Noirez P. Citrulline reduces glyceroneogenesis and induces fatty acid release in visceral adipose tissue from overweight rats. Mol Nutr Food Res. 2014 Dec;58(12):2320-30. doi: 10.1002/mnfr.201400507. Epub 2014 Oct 31. PMID 25271764
- [Background] Joffin N, Jaubert AM, Durant S, Bastin J, De Bandt JP, Cynober L, Moinard C, Forest C, Noirez P. Citrulline induces fatty acid release selectively in visceral adipose tissue from old rats. Mol Nutr Food Res. 2014 Sep;58(9):1765-75. doi: 10.1002/mnfr.201400053. Epub 2014 Jun 10. PMID 24913603
- [Background] Wu G, Collins JK, Perkins-Veazie P, Siddiq M, Dolan KD, Kelly KA, Heaps CL, Meininger CJ. Dietary supplementation with watermelon pomace juice enhances arginine availability and ameliorates the metabolic syndrome in Zucker diabetic fatty rats. J Nutr. 2007 Dec;137(12):2680-5. doi: 10.1093/jn/137.12.2680. PMID 18029483
- [Background] Morais JA, Chevalier S, Gougeon R. Protein turnover and requirements in the healthy and frail elderly. J Nutr Health Aging. 2006 Jul-Aug;10(4):272-83. PMID 16886097
- [Background] Skelton DA, Greig CA, Davies JM, Young A. Strength, power and related functional ability of healthy people aged 65-89 years. Age Ageing. 1994 Sep;23(5):371-7. doi: 10.1093/ageing/23.5.371. PMID 7825481
- [Background] Reid KF, Doros G, Clark DJ, Patten C, Carabello RJ, Cloutier GJ, Phillips EM, Krivickas LS, Frontera WR, Fielding RA. Muscle power failure in mobility-limited older adults: preserved single fiber function despite lower whole muscle size, quality and rate of neuromuscular activation. Eur J Appl Physiol. 2012 Jun;112(6):2289-301. doi: 10.1007/s00421-011-2200-0. Epub 2011 Oct 18. PMID 22005960
- [Background] Chen Z, Wang Z, Lohman T, Heymsfield SB, Outwater E, Nicholas JS, Bassford T, LaCroix A, Sherrill D, Punyanitya M, Wu G, Going S. Dual-energy X-ray absorptiometry is a valid tool for assessing skeletal muscle mass in older women. J Nutr. 2007 Dec;137(12):2775-80. doi: 10.1093/jn/137.12.2775. PMID 18029498
- [Background] Barbat-Artigas S, Rolland Y, Cesari M, Abellan van Kan G, Vellas B, Aubertin-Leheudre M. Clinical relevance of different muscle strength indexes and functional impairment in women aged 75 years and older. J Gerontol A Biol Sci Med Sci. 2013 Jul;68(7):811-9. doi: 10.1093/gerona/gls254. Epub 2012 Dec 21. PMID 23262030
- [Background] Jakicic JM, Marcus M, Gallagher KI, Randall C, Thomas E, Goss FL, Robertson RJ. Evaluation of the SenseWear Pro Armband to assess energy expenditure during exercise. Med Sci Sports Exerc. 2004 May;36(5):897-904. doi: 10.1249/01.mss.0000126805.32659.43. PMID 15126727
- [Background] Polzien KM, Jakicic JM, Tate DF, Otto AD. The efficacy of a technology-based system in a short-term behavioral weight loss intervention. Obesity (Silver Spring). 2007 Apr;15(4):825-30. doi: 10.1038/oby.2007.584. PMID 17426316
- [Background] Welk GJ, McClain JJ, Eisenmann JC, Wickel EE. Field validation of the MTI Actigraph and BodyMedia armband monitor using the IDEEA monitor. Obesity (Silver Spring). 2007 Apr;15(4):918-28. doi: 10.1038/oby.2007.624. PMID 17426327
- [Background] St-Onge M, Mignault D, Allison DB, Rabasa-Lhoret R. Evaluation of a portable device to measure daily energy expenditure in free-living adults. Am J Clin Nutr. 2007 Mar;85(3):742-9. doi: 10.1093/ajcn/85.3.742. PMID 17344495
- [Background] Luhrmann PM, Herbert BM, Gaster C, Neuhauser-Berthold M. Validation of a self-administered 3-day estimated dietary record for use in the elderly. Eur J Nutr. 1999 Oct;38(5):235-40. doi: 10.1007/s003940050066. PMID 10654160
- [Background] Chevalier S, Goulet ED, Burgos SA, Wykes LJ, Morais JA. Protein anabolic responses to a fed steady state in healthy aging. J Gerontol A Biol Sci Med Sci. 2011 Jun;66(6):681-8. doi: 10.1093/gerona/glr036. Epub 2011 Mar 24. PMID 21436253
- [Background] Gaudreau P, Morais JA, Shatenstein B, Gray-Donald K, Khalil A, Dionne I, Ferland G, Fulop T, Jacques D, Kergoat MJ, Tessier D, Wagner R, Payette H. Nutrition as a determinant of successful aging: description of the Quebec longitudinal study Nuage and results from cross-sectional pilot studies. Rejuvenation Res. 2007 Sep;10(3):377-86. doi: 10.1089/rej.2007.0596. PMID 17708689
- [Background] Yeap BB, Paul Chubb SA, Lopez D, Ho KK, Hankey GJ, Flicker L. Associations of insulin-like growth factor-I and its binding proteins and testosterone with frailty in older men. Clin Endocrinol (Oxf). 2013 May;78(5):752-9. doi: 10.1111/cen.12052. PMID 23009592
- [Background] Stephen WC, Janssen I. Sarcopenic-obesity and cardiovascular disease risk in the elderly. J Nutr Health Aging. 2009 May;13(5):460-6. doi: 10.1007/s12603-009-0084-z. PMID 19390754
- [Background] Braun MJ, Meta MD, Schneider P, Reiners C. Clinical evaluation of a high-resolution new peripheral quantitative computerized tomography (pQCT) scanner for the bone densitometry at the lower limbs. Phys Med Biol. 1998 Aug;43(8):2279-94. doi: 10.1088/0031-9155/43/8/020. PMID 9725604